CLINICAL TRIAL: NCT06993259
Title: Comparison of the Effectiveness of Virtual Reality and Serious Games on Pain, Fear, Anxiety, and Satisfaction During Skin Prick Testing in Children Aged 6-12 Years: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality and Serious Games on Pain, Fear, Anxiety, and Satisfaction During Skin Prick Testing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KOC_UNI
Record Dates: First submitted 2025-05-15; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pain; Anxiety; Fear; Allergy
MeSH Terms: conditions — Pain; Anxiety Disorders; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This research was designed as a randomized controlled trial with a parallel-group structure (intervention-control) to examine the effects of serious gaming and virtual reality interventions on reducing pain, fear, and anxiety levels, as well as improving care satisfaction among children aged 6-12 years who underwent skin prick tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention)
- Serious Game (Experimental)
  Interventions: Device: Serious game
- Virtual Reality (Experimental)
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Children in the virtual reality (VR) group watched a 360° Ice Age video via headset starting three minutes before and continuing throughout the allergy test. The video, selected by pediatric experts, was age-appropriate, visually rich, and emotionally neutral. VR provided immersive distraction to reduce pain, fear, and anxiety. After the test, children and parents rated pain (WBFPS), fear (CFS), anxiety (CAS-S), and satisfaction through structured forms.
  Arms: Virtual Reality
Device: Serious game — Children in the serious game group played Subway Surfers on a tablet starting three minutes before and continuing throughout the skin prick test. The game was chosen by pediatric experts for its age-appropriateness and ability to sustain attention without overstimulation. As a fast-paced, interactive tool, it served as an effective distraction to reduce pain, fear, and anxiety. After the procedure, children and parents rated pain (WBFPS), fear (CFS), anxiety (CAS-S), and satisfaction using structured feedback forms.
  Arms: Serious Game

SUMMARY:
This randomized controlled trial evaluated the effectiveness of virtual reality (VR) and serious gaming (SG) in reducing pain, fear, and anxiety, and improving satisfaction during skin prick testing (SPT) in children aged 6-12 years. A total of 90 children were randomly assigned to three groups: standard care (control), VR, or SG. The VR group watched a 360° animated video using a headset, while the SG group played Subway Surfers on a tablet. Pain (WBFPS), fear (CFS), anxiety (CAS-S), and satisfaction (VAS) were measured post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* Scheduled to undergo an allergy skin prick test
* No visual impairments
* No use of anxiolytic or analgesic medication within the past six hours
* Voluntary agreement to participate (child assent and parental consent)

Exclusion Criteria:

* Not within the 6-12 age range
* Not scheduled for an allergy skin prick test
* Presence of visual impairments
* Use of anxiolytic or analgesic medication within the past six hours
* Refusal to participate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale | Immediately after the skin prick test procedure (within 1-2 minutes post-intervention)
  The Wong-Baker FACES scale includes six facial expressions scored from 0 ("No Pain") to 10 ("Worst Pain"). Children select the face that best represents their pain. Valid for ages 3-18, it is widely used for its simplicity and strong psychometric properties and has been translated into many languages, including Turkish.
Child Fear Scale | Immediately after the skin prick test procedure (within 1-2 minutes post-intervention)
  The Child Fear Scale consists of six facial expressions scored from 0 (no fear) to 10 (highest fear) in increments of two. Fear increases progressively across the faces. Its validity and reliability were confirmed by Avşan et al. (2024), and it aligns with pain scales in format and scoring.
Child Anxiety State Scale | Immediately after the skin prick test procedure (within 1-2 minutes post-intervention)
  The Child Anxiety State Scale (CAS-S), developed by Ersig et al. (2013), was validated in Turkish by Özalp Gerçeker et al. (2019). Designed for children aged 4-10, it resembles a thermometer and measures current anxiety ("right now"). The scale has strong psychometric properties and is suitable for clinical use.

SECONDARY OUTCOMES:
VAS Care Satisfaction Score | Immediately after the skin prick test procedure (within 1-2 minutes post-intervention)
  The Visual Analog Scale (VAS) for care satisfaction was used to evaluate children's satisfaction with the care received during the allergy testing procedure. Children were asked to indicate their level of satisfaction on a scale ranging from "0 - Not satisfied at all" to "10 - Very satisfied."

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the lack of participant consent for data sharing beyond the scope of this study.